CLINICAL TRIAL: NCT03963570
Title: The Effectiveness of a Self-managed Digital Exercise Programme to Prevent Falls in Older Community-dwelling People -The Safe Step Randomized Controlled Trial
Brief Title: The Effectiveness of a Self-managed Digital Exercise Programme to Prevent Falls in Older Community-dwelling People
Acronym: SafeStepRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SafeStepRCT
Record Dates: First submitted 2019-04-15; First posted 2019-05-24 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Accidental Falls
Keywords: Accidental Falls; Prevention and control; Exercise; Exercise therapy/methods*; Aged; Aged 80 and over; Smartphone; Computers handheld; Motivation; Behaviour change; Postural balance; Health behaviour; mHealth; eHealth; Digital health; Self-management
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial (RCT) comparing a digital exercise program with a control group. The intervention will last for 12 months with follow-up assessments at 3, 6, 9 and 12 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All outcomes are self-reports and self-assessments by the participants and reported in digital surveys. Outcomes will not be influenced by any other outcome assessors. Data set will be blinded regarding group allocation (and the code for the groups will be held by a researcher not involved in the study) when performing analyses for main outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe Step - digital exercise program (Experimental): Participants randomized to the experimental group will receive full access to the Safe Step application and create their own individual program of strength and balance exercises. During 1 year the participants are recommended to exercise at least 30 minutes, 3 times a week and continuously progress their program. In addition they will every month receive an email with general falls prevention information in a short video.
  Interventions: Behavioral: Safe Step - digital exercise program
- Control group (Other): During 1 year, the participants randomized to the control group will receive an email every month with general falls prevention information in a short video.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Safe Step - digital exercise program — After receiving the Safe Step application the participants view an instruction movie on how to use the application to create and progress their own individual exercise program. The exercises, presented in video format, are organized into 10 predetermined groups with a main focus to improve balance (3 groups), increase lower-limb strength (4 groups), and improve gait/step (3 groups). The participants choose an exercise suitable for their needs from each group to compose a program of ten exercises.
  They can use the app to plan their exercises, set reminders, register their exercise, and view statistics of their progress. A virtual physiotherapist deliver motivational messages and feed-back. At the end of every month, of the 1 year intervention period, the participants will receive an email asking them to report any falls during the past month by answering a short digital survey. This message will provide a new video each month with general falls prevention information besides exercise.
  Arms: Safe Step - digital exercise program
Behavioral: Control group — Participants randomized to the control condition will only be given information. They will receive exactly the same email messages as the intervention group with falls prevention information and a request to report any falls. At the end of the 12 month intervention we will, in addition to the other questions, ask if they have started to do any exercises during the intervention period. After the 12 month follow-up assessment the control group will be offered the Safe Step application.
  Arms: Control group

SUMMARY:
The overall aim of the study is to evaluate the effectiveness of a digital self-management exercise program in preventing falls in community dwelling older people.

Participants will be recruited in Sweden through the website (www.sakrasteg.se) providing study information. On the website interested seniors will get information about the aim and procedures of the study as well as inclusion and exclusion criteria. If seniors themselves judge that they are eligible to participate in the study they can register by providing their email address. After baseline assessment, through self-reports in a digital survey, participants will be randomized to either an exercise intervention or a control group in a 1:1 ratio. The investigators aim to include 1400 participants and recruitment will be ongoing continuously for one year.

The exercise intervention is delivered through the Safe Step application, developed in co-creation with seniors and an interdisciplinary research team. Safe Step provides a large repository of evidence based exercises in video formats alongside falls preventive information and advice. With support of this application the user can compose an individualized exercise program with balance and strength exercises suitable for their needs. To help the user adhere to the program a set of behaviour change techniques is provided by the program. The user can set their own goals, get reminders and positive feedback form a virtual physiotherapist, and follow their own progress. Advice on how to integrate the exercises into everyday activities is also offered. The participants will exercise on their own with the help of the application during one year, with a recommendation of 30 minutes at least 3 times/week.

In addition to the exercise intervention the participants will every month get an email with falls preventive information in short videos, they will also be asked to report any falls by responding to a survey attached to the message. The exercise group will be compared to a control group that will receive the same information emails as the exercise group, but no individual exercise advice.

The interventions will last for 1 year with follow up assessments at 3, 6, 9, and 12 month in addition the monthly fall reports. Due to the nature of the study, with no face to face contact, all outcome measures are self-reports and self-tests in digital surveys. The primary outcome is fall rate. The study follows the CONSORT guidelines and CONSORT EHEALTH criteria.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older
* Have fallen or experienced a decline in perceived postural balance during the last year
* Have access to a smartphone or a tablet and uses it regularly
* Have an own email address and uses it
* Ability to understand verbal and written instructions in Swedish
* Can rise from a standard height chair without a person helping
* Independently mobile without a walking aid indoors

Exclusion Criteria:

* Progressive disease where there is likely to be a decline in strength or balance over the next year
* Perceived memory dysfunction that affect everyday life activities
* Taking part in more than 3 hours each week of strenuous physical exercise which makes them out of breath (e.g. dance, gymnastics, gym exercises, running or skiing)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1628 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Fall rate | 12 months
  Falls will be registered every month through a short digital survey, received by email, asking the participant if they had any falls during the last month. If answering yes a few additional questions about when the fall occurred, any resulting injuries and hospital visits will be asked.

SECONDARY OUTCOMES:
Functional leg strength | Change; Baseline, 3 months, 6 months, 9 months, 12 months
  Self-administered chair stand test (i.e. number of stands during 30 seconds).
Perceived Exertion | Change; Baseline, 3 months, 6 months, 9 months, 12 months
  The Borg Scale of Perceived Exertion during the 30 second chair stand test, rated on a scale between 6 (none) to 20 (maximal exertion).
Self-rated balance | Change; Baseline, 3 months, 6 months, 9 months, 12 months
  Answering the question: "How do you perceive you balance?" on a 5-level ordinal scale ranging from "very good" to "very bad".
Self-rated leg-strength | Change; Baseline, 3 months, 6 months, 9 months, 12 months
  Answering the question: "How do you perceive your leg muscle strength?" on a 5-level ordinal scale ranging from "very good" to "very bad".
Falls efficacy | Change; Baseline, 3 months, 6 months, 9 months, 12 months
  Falls Efficacy Scale-International (FES-I). Concerns about falling is rated for 16 activities (e.g. cleaning the house) on a scale from 1 (not at all concerned ) to 4 (very concerned ). Ratings for each of the 16 activities are summed to a total score ranging from 16 (no concern about falling) to maximum 64 (severe concern about falling)
Health related quality of life | Change; Baseline, 3 months, 6 months, 9 months, 12 months
  Health related quality of life is assessed by the EuroQol 5 dimension 5 level self-report questionnaire (EQ-5D-5L).
  The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and a Visual Analogue scale (VAS). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. A 1-digit number express the level selected for each dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. It should be noted that the numerals 1-5 have no arithmetic properties. The VAS records the respondent's self-rated health on a vertical, visual analogue scale (ranging from 0-100) with endpoints labelled "the best health you can imagine" and "the worst health you can imagine".
  .
Use of the information videos | 3 months, 6 months, 9 months, 12 months
  Answering the question: "Have you watched the videos we sent you by e-mail during the last 3 months?" on a 4-level ordinal scale.
Experienced positive effects of the exercise intervention | 3 months, 6 months, 9 months, 12 months
  Exercise intervention: Self-report of any positive effects of the exercise intervention besides effects on balance and strength. On a nominal scale including an optional text field.
Experienced negative effects of the exercise intervention | 3 months, 6 months, 9 months, 12 months
  Exercise intervention: Self-report of any negative effects (adverse events) of the exercise intervention besides effects on balance and strength. On a nominal scale including an optional text field.
Physical activity | Change: Baseline, 12 months
  Self-reported minutes/week, pre-defined alternatives in 30 minutes blocks up to more than 2 hours.
Number of fallers | 12 months
  Falls will be registered every month through a short digital survey, received by email, asking the participant if they had any falls during the last month. If answering yes a few additional questions about when the fall occurred, any resulting injuries and hospital visits will be asked.
Exercise adherence throughout the intervention | 12 months
  Exercise intervention: Adherence to predefined minutes of 3x30 min/week reported continuously through an integrated exercise diary in the Safe step application and by self-report at follow up assessments.
Self-rated improvements in balance | 12 months
  Answering the question: "If you compare with when you started this study a year ago, how would you assess balance today?" on a 5-level ordinal scale on a 5-level ordinal scale ranging from "much better" to "much worse".
Self-rated improvements in leg-strength | 12 months
  Answering the questions: "If you compare with when you started this study a year ago, how would you assess the muscle strength in your legs today?" on a 5-level ordinal scale ranging from "much better" to "much worse".
Rate of attrition | 12 months
  Drop-outs and with-draws in the study
Sociodemographic characteristics | Baseline
  Reach of recruitment will be assessed based on self-reported sociodemographic characteristics of participants included.
New exercise routines | 12 months
  Participants will be asked if they have started to do any exercises (besides the study intervention) during the intervention period.
Costs related to the interventions | 12 months
  Participants will be asked to report if they have had any cost related to the intervention during the intervention period e.g. for internet access or equipment.
Cost-effectiveness | 12 months
  Cost-effectiveness of the interventions with respect to falls

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Sandlund, Assist. Prof, Principal Investigator — Umeå University
Locations (1):
- Caring Science Buildning, Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: Will be published October-November 2019
Access Criteria: Data will be available from the corresponding author on reasonable request. The protocol will be published in an open access journal.

REFERENCES:
- [Derived] Pettersson B, Lundin-Olsson L, Skelton DA, Liv P, Zingmark M, Rosendahl E, Sandlund M. Effectiveness of the Safe Step Digital Exercise Program to Prevent Falls in Older Community-Dwelling Adults: Randomized Controlled Trial. J Med Internet Res. 2025 Mar 31;27:e67539. doi: 10.2196/67539. PMID 40163860
- [Derived] Pettersson B, Lundin-Olsson L, Skelton DA, Liv P, Zingmark M, Rosendahl E, Sandlund M. Effectiveness of a self-managed digital exercise programme to prevent falls in older community-dwelling adults: study protocol for the Safe Step randomised controlled trial. BMJ Open. 2020 May 17;10(5):e036194. doi: 10.1136/bmjopen-2019-036194. PMID 32423936
- See also: Project web-site — http://www.sakrasteg.se